CLINICAL TRIAL: NCT06017115
Title: Evaluation of Straumann Bone Level Tapered® Implants Using Screwed Abutment Height in Partially Edentulous Patients: a Randomized Controlled Clinical Trial
Brief Title: Evaluation of Using Different Screwed Abutment Height
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jordi Gargallo-Albiol, Associate Professor of Oral and Maxillofacial Surgery, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIR-ECL-2016-03
Record Dates: First submitted 2023-06-29; First posted 2023-08-30 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Bone Loss
Keywords: bone loss; dental implant; bone implant interface; Peri implant Endosseous Healing; Dental implant abutment
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Each patient will be randomly allocated in one of the two groups: test group (n=36) or control group (n=12)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Group 1: 2 stage approach (cover screw) (12 patients): cover screw is placed over the dental implants in the first surgery and a second surgery will be performed to expose the implants and placing a healing abutment after 2-4 months, DEVICES: COVER SCREW (first surgery) and HEALING ABUTMENT (second surgery)
  Interventions: Device: Dental implant placement with COVER SCREW (two surgeries in control group) or DEFINITIVE TRANSEPITHELIAL ABUTMENT (one surgery in test group)
- Test group (Experimental): Group 2: Protective plastic cap over different definitive trans-epithelial abutments are placed in the unic surgery performed (36 patients): Definitive transepithelial abutments will be placed the same day of the implant placement surgery. DEVICE: DEFINITIVE TRANSEPITHELIAL ABUTMENT
  Interventions: Device: Dental implant placement with COVER SCREW (two surgeries in control group) or DEFINITIVE TRANSEPITHELIAL ABUTMENT (one surgery in test group)

INTERVENTIONS:
Device: Dental implant placement with COVER SCREW (two surgeries in control group) or DEFINITIVE TRANSEPITHELIAL ABUTMENT (one surgery in test group) — Dental implant placement using cover screws (first surgery) and a healing abutment (second surgery) or definitive transepithelial abutments the same day of the implant placement (one unit surgery)

SUMMARY:
A prospective randomized controlled clinical trial will be conducted. Study groups will be assigned as described above. The patients will be randomly divided into two groups in order to study the influence of prosthetic screw abutment in marginal bone loss (MBL) around Bone Level Tapered implants (BLT® Roxolid® SLActive® guided implants, Straumann Dental Implant System, Institut Straumann AG, Basel, Switzerland).

DETAILED DESCRIPTION:
48 patients will be selected with partial edentulism in the maxilla or mandible, requiring two dental implants in the posterior areas (molars and premolars).

Each patient will be randomly allocated in one of the two groups: test group (n=36) or control group (n=12) and all the implants will be placed by residents of the International Master in Oral Surgery and Master in Periodontics of the same University.

Study groups

Group 1: Two stage approach (cover screw in first surgery and healing abutment in second surgery) (12 patients)

Group 2: One stage approach (healing cap over trans-epithelial abutments) (36 patients).Two subgroups according to different trans-epithelial height abutment:

* Subgroup 2.1: Screw-retained abutment of 1 mm height (18 patients)
* Subgroup 2.2: Screw-retained abutment of 2.5 mm height (18 patients)

Clinical Parameters and Outcomes

* Three-dimensional volumetric changes in hard and soft tissues (Cone-beam computed tomography superposed with digital cast models).
* Marginal bone level (MBL) change: Standardized intraoral periapical x-rays will be taken on the day of surgery, 4, 6, 12, 24 and 36 months following surgery.
* Probing depth, bleeding on probing and keratinized mucosa width will be measured in the follow-up visits in 3 different points in buccal (Mesial, center and distal).
* VAS Scale: The visual analog scale or visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Overall, healthy subjects
3. Females and males of at least eighteen-years
4. Requiring a minimum of two implants (molar and/or premolar teeth)
5. Adequate oral hygiene (less than 15% FMPS)
6. Able to follow instructions and attend a regular compliance
7. Enough bone to place a standard implant of 4.1 mm diameter.

Exclusion Criteria:

1. Acute local infection
2. Occlusal overload with parafunctional activity (assessed clinically)
3. Large occlusal discrepancies
4. Untreated periodontal disease assessed by Socransky et al. parameters (≥2mm clinical attachment loss in two consecutive visits within 1 year)
5. Smokers (more than 10 cigarettes/day)
6. Drug and/or alcoholic dependencies
7. Medical conditions contraindicating implant surgery
8. History of head and/or neck radiation
9. Bisphosphonate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Gargallo-Albiol, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The investigators will have all the informed consent forms, the clinical study report, the presurgical plan, the CBCT immediately post-surgery, and the outcome variable tables of each follow-up visit.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The first outcome will be available in July-2022 and the last outcome in July.2024

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: implant
Period: Overall Study
Arm/Group | Control Group | Test Group
Started | 12; 24 implant | 18; 36 implant
Completed | 12; 24 implant | 18; 36 implant
Not Completed | 0; 0 implant | 0; 0 implant

BASELINE CHARACTERISTICS:
Population: A total of 30 patients (12 of the control group and 18 of the test group) started the study and complete the 24 months of follow-up.
Units Other Than Participants: implant
Groups:
- Control Group: Two Stage Approach: Implant placement surgery with close screw and sumerge implant approach
- Test Group: One Stage Approach: Implant placement surgery with trans-epithelial abutment
- Total: Total of all reporting groups
Arm/Group | Control Group: Two Stage Approach | Test Group: One Stage Approach | Total
Number analyzed (Participants) | 12 | 18 | 30
Number analyzed (implant) | 24 | 36 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.90 (9.09) | 63.28 (9.79) | 65.77 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 9 | 12 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Marginal bone loss [Mean (Standard Deviation); unit: millimeters] | 1.17 (0.36) | 0.83 (0.26) | 0.97 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Loss
Description: Periimplant bone level by measuring from the implant platform to the first bone to implant contact. Messuret in 2 points: MESIAL AND DISTAL with intra-oral XR. (measured in millimeters). The mean of this two-points for each implant was calculated. Afterwards, the mean for the mesial implants, distal and total implant sample per group was calculated.
Time Frame: After implant loading (baseline)and once every year to 24 months follow-up
Population: A total of 30 patients (60 implants), 12 of the control group (24 implants) and 18 of the test group (36 implants) were assessed after 24 months follow-up.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: implants
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 12 | 18
Number analyzed (implants) | 24 | 36
millimeters
  Total implants at 24 months | 1.17 (0.35) | 0.83 (0.25)
  Mesial implant at 24 months | 1.28 (0.47) | 0.96 (0.36)
  Distal implant at 24 months | 1.06 (0.53) | 0.71 (0.27)
  Total implants at 12 months | 1.13 (0.34) | 0.80 (0.26)
  Mesial implant at 12 months | 1.25 (0.46) | 0.93 (0.38)
  Distal implant at 12 months | 0.81 (0.41) | 0.67 (0.27)

2. Secondary Outcome: Probing Depth
Description: Measuring this outcomes at 4 different points .(Mesial Buccal, Center Buccal, Distal Buccal and central lingual) (measured in millimeters).
Time Frame: After implant loading (baseline)and once every year to 36 months follow-up
Reporting Status: Not Posted

3. Secondary Outcome: Bleeding on Probing
Description: as for outcome 2
Time Frame: After implant loading (baseline)and once every year to 36 months follow-up
Reporting Status: Not Posted

4. Secondary Outcome: Keratinized Mucosa Width
Description: as for outcome 2
Time Frame: After implant loading (baseline)and once every year to 36 months follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Control Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 0/12 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT06017115/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT06017115/SAP_001.pdf
  • Informed Consent Form (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT06017115/ICF_002.pdf